CLINICAL TRIAL: NCT04817020
Title: Effect of Skin Antisepsis on Phlebitis in Peripheral Intravenous Catheter
Brief Title: Effect of Skin Antisepsis on Phlebitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Alev Keskin, Principle investigator, Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: AKeskin
Record Dates: First submitted 2021-03-19; First posted 2021-03-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Phlebitis
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Intervention Model Description: Randomize,controlled double-blind clinical trials
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Klorheksidin (Experimental): Deri antisepsisi, vasküler erişimden önce chlorhexidine kullanılarak yapılacaktır
  Interventions: Other: %2 Klorheksidin
- Alkol (Experimental): Skin antisepsis will be performed using alcohol prior to vascular access
  Interventions: Other: %2 Klorheksidin

INTERVENTIONS:
Other: %2 Klorheksidin — Effect on phlebitis
  Other Names: % 70 Alchol

SUMMARY:
Peripheral intravenous catheters have application such as fluid, blood, medication and feding fluids. Although it is a life-savingtool, it can lead to some complications as a result of incorrect applications. Phlebitis, which is defined as inflammation of the tunica intima layer of the vein, is characterized by pain, redness, tenderness, palpable stiffness and increased temperature. As can be seen during catheter application, it can develop within 48-96 hours after catheter removal. Instudies performed, the rate of phlebitis development was 0.1-63.3% in patients with peripheral intravenous catheters, in Turkey, this rate varies between 11% and 67%.

Phlebitis; can be originated mechanical, chemical and bacterial. Various guidelines are available from evidence based on research results to prevent and reduce phlebitis development. In our country, National Vascular Access Management Guide is used.

One of the principles in the National Guidelines for Vascular Access Management for the prevention of phlebitis is skin antisepsis. The guideline recommends a 70% alcohol solution containing>0.5% chlorhexidine for skin antisepsis and reports that povidone-iodine or only 70% alcohol solution can be used in the absence or contraindication. Infusion Nurses Society (INS, 2016) recommends using the 'Phlebitis Scale' in the early diagnosis of phlebitis.

In this study, investigator aimed to compare the antiseptic effects of 2% chlorhexidine and 70% alcohol which are used as antiseptic in preventing phlebitis development while providing skin antisepsis, which is one of the basic principles in the application of peripheral intravenous catheter. This study is a randomized controlled clinical study and the population will consist of patients (participants)hospitalized in the Surgery -1 Department of Balcalı Hospital, Faculty of Medicine, Çukurova University.

As a data collection tool; 'Patient Information Form' and 'İnformation Form for İntravenous Catheter Application to the Patient' created by there searcher, to evaluate phlebitis formation "Phlebitis Scale'' which published by the Infusion Nurses Society (INS, 2016) will be used. A transparent millimeter ruler will be used

DETAILED DESCRIPTION:
In the study, data were collected for 9 months between January 2020 and September 2020.

Before starting the research, the nurses in the clinic were informed about the work to be done. Participants who were admitted to the surgical service, who met the inclusion criteria and accepted to participate in the study on a voluntary basis were separated into two groups by block randomization method. Then, the participants assigned to the groups were informed about the study and the "Patient Information Form" was administered by the researcher after obtaining the consent of the individuals.

In order to eliminate the bias regarding the antiseptic used while inserting the catheter, investigator did not have information about the solution used, participants and nurses in the clinic. The solutions were prepared by the nurse in charge of the Surgery 1 Clinic. Both solutions were put into bottles of the same color and size. It was a light proof bottle in both bottles. The usage dates of both solutions were checked. As they were transferred to different bottles, the bottles and solutions were renewed once a month by the nurse in charge with the recommendation of the hospital infection control committee. A pink sticker was attached to one of the bottles (to cover the entire bottle), and a blue sticker to the other (to cover the entire bottle). Which color and which solution was known only by the clinic responsible nurses.

As stated in the statement of the nurse in charge of the surgery 1 service, he wrote the color which solution was on a piece of paper and put it in a sealed envelope. D He prepared two of the same envelopes and gave the other one to the responsible nurse of the General Surgery-2 Clinic. The envelopes were kept by both responsible until the end of the work. Solutions could not be distinguished in terms of color and odor. After the study comes from statistics, when looking at the solutions by opening the closed envelope; It was observed that 2% chlorhexidine was used in the participants in group 1 (blue solution) selected by randomization method, and 70% alcohol was used in the second group (pink solution) by investigator.İ.V. A sterile, transparent, semi-permeable, self-adhesive catheter stabilizer was used as a catheter cover for all patients in Group 1 and Group 2. İ.V. After catheterization, "Information Form Regarding IV Catheter Application to Patient" was filled in for each participant.

Desefin and (active substance: ceftriaxone) biteral (active substance: ornidazole) and parol (active substance: paracetamol) as an analgesic were administered through the intravenous catheter inserted for the study. It was ensured that these drugs were sent in the form of infusion. Therefore, verbal consent was obtained from the participants to apply the catheter for the second time, except for the intravenous catheter attached, if the patient was to receive different intravenous therapy.

After the application, phlebitis development status was evaluated with the "Phlebitis Scale" published by the Infusion Nurses Association. As part of the follow-up of phlebitis, millimetric measurements were made with a transparent ruler and the degree of phlebitis was determined bu intestigator. The scale was applied every 8 hours for 72 hours by investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65, Patients who accept the study,

  * Patients newly admitted to the clinic,
  * Patients whose vascular access will be opened in the clinic,
  * Patients whose upper extremity can be used for vascular access, Patients not receiving chemotherapy, Patients using antibiotics and analgesics containing the same active substance in intravenous drug treatment, Patients not discharged before 72 hours,
  * Patients without blood disease, Patients without peripheral vascular disease,

Exclusion Criteria:

Patients younger than 18 and older than 65, Patients who do not accept the study, Patients with peripheral vascular disease, Patients with blood disease, Patients receiving chemotherapy,

* Patients who do not use the upper extremity,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-10-16 (Actual)

PRIMARY OUTCOMES:
Patient information form | 5 minute
  The "Patient Information Form" created by the researcher using the literature consists of 15 questions. Demographic information of the patient (diagnosis, age, gender, weight, height, body mass index, chronic disease, alcohol, smoking, allergy, edema in hands and feet) and intravenous drugs and these drugs It consists of questions that give information about how it is done.
Information Form Regarding the Application of the IV Catheter to the Patient | 30 minute
  In the form created by the researcher by scanning the literature, the date and time of the intravenous catheter insertion and removal, the size of the catheter, the area where the catheter was inserted, the number of trials the catheter was inserted, and the precaution package to be applied during catheter insertion published by the National Vascular Access Management Guide (2019) There are questions created by using the catheter, guiding the person wearing the catheter and giving information about what kind of antisepsis was performed during the insertion of the catheter.
Phlebitis Scale | 72 hours
  The phlebitis scale developed by the Infusion Nurses Society (INS, 2006) and recommended for use all over the world was used to determine the development status and degree of phlebitis.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Çukurova üniversitesi sağlık bilimleri fakültesi, Adana, Sarıçam
  - Çukurova university, Adana